CLINICAL TRIAL: NCT00774072
Title: Nasal Inhalation of Tobramycin by the Pari Sinus Nebulizer in Patients With Cystic Fibrosis and Pseudomonas Aeruginosa Colonization in the Upper Airways
Brief Title: Nasal Inhalation of Tobramycin in Patients With Cystic Fibrosis and Pseudomonas Aeruginosa Colonization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, PD Dr. Jochen G. Mainz, Head, CF Center, University of Jena
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: tobra nasal CF pilot
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Cystic Fibrosis; Pseudomonas Aeruginosa
Keywords: subjects with cystic fibrosis and pseudomonas aeruginosa colonization in the upper airways
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — Tobramycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tobramycin 80 mg (Active Comparator): applied once daily via Pari Sinus nebulizer
  Interventions: Drug: Tobramycin (Gernebcin®)
- isotonic saline (Placebo Comparator): applied once daily via Pari Sinus nebulizer
  Interventions: Drug: Tobramycin (Gernebcin®)

INTERVENTIONS:
Drug: Tobramycin (Gernebcin®) — 1 ml / day in each nostril

SUMMARY:
The purpose of this study is to determine whether the nasal inhalation of Gernebcin® is effective to decrease the Pseudomonas aeruginosa bacterial count in the nasal lavage fluid.

ELIGIBILITY:
Inclusion Criteria:

* subject has a confirmed diagnosis of cystic fibrosis
* detection of P. aeruginosa in nasal lavage (culture) with chronic P.a. colonization of the lung (from day -28)
* informed consent of the patients or parents
* subject is older than 7 years
* subject is able to comply with the inhalation procedures and nasal lavage procedures scheduled in the protocol
* women of childbearing potential are only included into the study, if they are using an effective method of birth control during the protocol

Exclusion Criteria:

* subject has a critical condition defined as: FEV1 < 30% and / or SaO2 < 93% without O2-substitution; need of O2-substitution
* subject had an ENT surgery within 3 months prior to study
* subject shows signs of nasal bleeding
* subject has an ear drum perforation
* subject had an acute rhinosinusitis or a pulmonary exacerbation at study entry with need of additional systemic antibiotic therapy against pseudomonas aerug.
* subject is unlikely to comply with the procedures scheduled in the protocol
* subject has a known allergic reaction to the medication
* subject is pregnant or breastfeeding
* subject participates in another clinical trial within 30 days prior to study entry or 30 days after end of the study.
* systemic (oral or intravenous) antibiotic treatment against P.a. 14 days prior to the inclusion and during the study
* if serum level of tobramycin is above 2 mg/l one hour after inhalation, subject has to withdraw the participation in the study.
* progressed renal insufficiency
* severe damage of the N. acusticus
* dizziness (potential damage of. N. vestibularis)

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Decrease of Pseudomonas aeruginosa bacterial count in the nasal lavage fluid | day -1, 1, 29, 30, 59, 60

SECONDARY OUTCOMES:
Measure of serum levels of tobramycin | day 1, 30 and 60
Tolerability | day 1, 30 and 60

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Mainz, M.D., Study Chair — University of Jena, Children's hospital
Locations (2):
- Germany (2):
  - Universitäts-Kinderklinik, Tübingen, Baden-Würtemberg
  - Mukoviszidosezentrum der Friedrich-Schiller-Universität, Jena, Thuringia

REFERENCES:
- [Background] Mainz JG, Arnold C. Authors' reply. Drug Des Devel Ther. 2014;8:1136-7. No abstract available. PMID 25199217
- [Background] Mainz JG, Michl R, Pfister W, Beck JF. Cystic fibrosis upper airways primary colonization with Pseudomonas aeruginosa: eradicated by sinonasal antibiotic inhalation. Am J Respir Crit Care Med. 2011 Nov 1;184(9):1089-90. doi: 10.1164/ajrccm.184.9.1089. No abstract available. PMID 22045752
- [Result] Mainz JG, Schadlich K, Schien C, Michl R, Schelhorn-Neise P, Koitschev A, Koitschev C, Keller PM, Riethmuller J, Wiedemann B, Beck JF. Sinonasal inhalation of tobramycin vibrating aerosol in cystic fibrosis patients with upper airway Pseudomonas aeruginosa colonization: results of a randomized, double-blind, placebo-controlled pilot study. Drug Des Devel Ther. 2014 Feb 10;8:209-17. doi: 10.2147/DDDT.S54064. eCollection 2014. PMID 24596456